CLINICAL TRIAL: NCT05172765
Title: Biomarker-Guided Optimization of Transcutaneous Vagal Stimulation for Atrial (BiG tVNS-AF)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 13786
Record Dates: First submitted 2021-10-21; First posted 2021-12-29 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active TENS Stimulation (Active Comparator)
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation Device
- Inactive TENS Stimulation (Sham Comparator)
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation Device

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation Device — Low-level, electrical stimulation of the outer ear (LLTS), using a transcutaneous electrical nerve stimulation (TENS) device.

SUMMARY:
This proposal aims to determine the effects of tVNS on autonomic tone, atrial substrate and neuromodulators in patients with paroxysmal atrial fibrillation (AF), investigate the chronic effects of optimal tVNS on AF burden in patients with paroxysmal AF over a 6-month period, compared with sham stimulation, and identify physiological and biochemical markers of response to chronic tVNS.

DETAILED DESCRIPTION:
This proposal aims to 1. To determine the effects of tVNS on autonomic tone, atrial substrate and neuromodulators in patients with paroxysmal atrial fibrillation (AF), 2. Investigate the chronic effects of optimal tVNS on AF burden in patients with paroxysmal AF over a 6-month period, compared with sham stimulation, and 3. To identify physiological and biochemical markers of response to chronic tVNS. For Aim 1, patients with paroxysmal AF will be randomized to a series of stimulation frequencies (5Hz, 10Hz, 20Hz) and intensities (50% below, and 1mA lower than, the discomfort threshold, respectively) in a cross-over design, to define optimal effects and 'dosing' of tVNS. Heart rate variability, a marker of autonomic tone and PWA, will be derived from 5-minute ECG. A subgroup of these patients, who present to the Electrophysiology laboratory for AF ablation, will be randomized to active or sham tVNS, using the optimal parameters determined above, for 5 minutes prior to any ablation, under baseline conditions, during isoproterenol or atropine infusion, and their combination. PWA will be estimated based on a 5-min ECG. The level of NPY will be measured from peripheral vein and coronary sinus samples. In this this Aim we will determine the optimal parameters for tVNS, and if the response to tVNS is dependent on the underlying autonomic tone. For Aim 2, Patients with paroxysmal AF not undergoing ablation, will be randomized to active tVNS (1 hour or 30 minutes, daily) or sham tVNS (1 hour daily) for 6 months, using the optimal tVNS parameters determined in Aim 1. AF burden will be monitored continuously using a smartwatch. In addition, all patients will receive a short trial of acute tVNS at baseline. This Aim will determine the minimum duration of tVNS needed to achieve a decrease in AF burden. Patients participating in the clinical trial described in Aim 2, will comprise the population of Aim 3. The hypothesis is that patients who respond acutely to tVNS at baseline, as assessed by PWA, are more likely to benefit from chronic tVNS therapy. Blood samples will be collected from patients participating in Aim 2, and their NPY levels and metabolomic profile will be correlated with AF burden. The results of these studies will first, provide insights into the effects of tVNS on autonomic tone, AF substrate and neuromodulators, and second, permit optimization of tVNS using PWA, NPY and metabolomic biomarkers to reduce AF burden of afflicted patients. By introducing an optimized tVNS treatment protocol, results from our proposed studies have the potential to overturn the current scientific paradigm for treatment of AF, and thus, lead to major improvements in health care delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Paroxysmal atrial fibrillation

Exclusion Criteria:

1. Sick sinus syndrome
2. 2nd and 3rd degree AV block (without pacemaker), bifascicular block or prolonged (PR>300ms) 1st degree AV block
3. History of vagotomy
4. Recurrent vasovagal syncope
5. Left ventricular ejection fraction < 40%
6. Significant valvular disorder (i.e., prosthetic valve or hemodynamic significant valvular diseases)
7. Recent stroke (< 3 months)
8. Myocardial infarction or hospitalization for heart failure (< 3 months)
9. Severe heart failure (NYHA Class IV)
10. End stage kidney disease on dialysis
11. Pregnancy

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-09-14 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
Effects of tVNS on Atrial fibrillation burden | 6 months
  AF burden, defined as the percent of time spent in AF over the total monitoring period, will be determined be based on continuous monitoring with an Apple watch

SECONDARY OUTCOMES:
Effects of tVNS on neuropeptide Y | 6 months
  Neuropeptide Y levels will be determined using commercially available ELISA kits
Effects of tVNS on Autonomic Tone | 6 months
  We will use heart rate variability (HRV) to assess the effect of tVNS on autonomic tone. HRV will be derived from a 5-minute ECG.
Effects of tVNS on P wave alternans | 6 months
  A 12-lead, high resolution ECG will be performed to determine P wave alternance, using a software that analyzes subtle beta-to-beat variations in P wave amplitude. The percentage of beats showing P wave alternans divided by the total number of beats represents P wave alternans burden.

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Stavrakis, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States